CLINICAL TRIAL: NCT03117894
Title: Regional Anesthesia for Breast Cancer Surgery, Effects on Postoperative Wellbeing and Disease Recurrence.
Brief Title: PECS-2 for Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UmeaU-PECS
Record Dates: First submitted 2017-03-06; First posted 2017-04-18 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Breast Neoplasm Female; Regional Anesthesia; Anesthesia; Regional Anesthesia Morbidity; Anesthesia Morbidity
MeSH Terms: interventions — Ropivacaine; Propofol; Etoricoxib; Ondansetron; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GA with RA (Active Comparator): Regional Anesthesia and General Anesthesia.
  Interventions: Drug: Ropivacaine 5 mg/ml, 35 ml; Drug: Remifentanil 50 microg/ml; Drug: Betamethason 4 mg; Drug: Paracetamol 1,5 g; Drug: Propofol; Drug: Arcoxia, 120 mg; Drug: Ondansetron 4 mg
- GA without RA (Active Comparator): Only General Anesthesia (without a supplemental Regional Anesthesia).
  Interventions: Drug: Remifentanil 50 microg/ml; Drug: Betamethason 4 mg; Drug: Paracetamol 1,5 g; Drug: Propofol; Drug: Arcoxia, 120 mg; Drug: Ondansetron 4 mg; Drug: Morphine

INTERVENTIONS:
Drug: Ropivacaine 5 mg/ml, 35 ml — Regional Anesthesia. The deposition of local anesthetics in proximity of nerves with the aim of blocking nerve transmission. This is used to block pain as an alternative to systemic treatment of pain.
  Arms: GA with RA
Drug: Remifentanil 50 microg/ml — The intravenous administration of anesthetics aiming to induce analgesia (part of the general anesthesia). No fixed dose, administered in relation to the study participants need at the moment.
Drug: Betamethason 4 mg — Are meant to decrease the risk of so called postoperative nausea and vomiting (PONV). Administered preoperatively.
Drug: Paracetamol 1,5 g — Administered preoperatively to prevent pain postoperatively.
  Other Names: Prevention of pain
Drug: Propofol — The intravenous administration of anesthetics aiming to induce sleep (part of the general anesthesia). No fixed dose, administered in relation to the study participants need at the moment.
Drug: Arcoxia, 120 mg — Administered preoperatively to prevent pain postoperatively.
Drug: Ondansetron 4 mg — Are meant to decrease the risk of so called postoperative nausea and vomiting (PONV). Administered peroperative.
Drug: Morphine — Administered peroperative, at the end of the surgery, before awakening the study participant. The aim is to prevent pain.
  Arms: GA without RA

SUMMARY:
There is no consensus regarding which alternative is the best anesthesia for breast surgery, general anesthesia and morphine for postoperative analgesia or a combination of regional anesthesia and general anesthesia that possibly attenuates or abolishes the need for morphine.

The current study aims to determine which of the two strategies that is best in relation to postoperative pain, nausea and risk of recurrence of the disease.

DETAILED DESCRIPTION:
Surgery for suspected or confirmed breast cancer is a common procedure world wide. The Swedish National board of health- and welfare reports that > 7000 women is diagnosed with breast cancer each year in Sweden.

Surgery always comes at the cost of a painful stimuli. It is of great importance that the anesthetist has anticipated this pain and has a plan to handle it.

The most common way to do this is to anesthetise the patient (put him or her to sleep, also called a General Anesthesia (GA)) for the surgical procedure and administer a strong analgesic (usually morphine) before the patient is awaken. Morphine has side-effects.

Another possible plan is to rely on a Regional Anesthesia (RA) (block pain from a certain part of the body) to take care of the pain, both during and after the surgery. Thereby this patient may be awake during the surgery. The two strategies may also be combined. That is, a regional anesthesia is applied before surgery but the patient is also put to sleep. The regional anesthesia is then fully effective when the patient is awaken and no strong analgesics are administered. The approach with a regional anesthesia is common in orthopedic surgery, either in combination with or without a general anesthesia.

For surgery on the breast, there has been few alternatives available for regional anesthesia. They have been considered to invasive for regular use and not been incorporated in clinical praxis as a routine.

The praxis of regional anesthesia has expanded tremendously in recent years. This is attributed to the increased use of ultrasound as a guide for the injection of anesthetic compounds in proximity to the nerves. The pectoral nerve block (PECS) was first described in 2011. It has since then been developed further and is much more feasible than the older alternatives for regional anesthesia covering the breast.

Therefore it has gained some popularity and a few studies on its performance have been published in recent years. It is still not clear though, if it really confers the patient a better postoperative situation regarding pain and nausea.

Further, observational studies have suggested that malignant disease is spread and hence recurs less often if the surgery is performed in conjunction with a regional anesthesia. These results have not yet been confirmed in randomized trials. Therefore, the investigators will use the data from the current study and also look if there is a difference between the study groups regarding recurrence of the disease and mortality three and five years after inclusion in the study.

A subgroup analysis will be made on the patients that has a mastectomy.

ELIGIBILITY:
Inclusion Criteria: Unilateral surgery on the breast because of suspected malign disease.

Exclusion Criteria:

Bilateral surgery

Metastases other than in the axilla

Body Mass Index (BMI) > 35

Not able to communicate in Swedish

Dementia

American Society of Anesthesiology (ASA) 4 or 5

Chronic pain treatment (use of opiates or medicine for neuropathic pain > 7 days the last month)

Known allergy to Morphine or Ropivacaine

Congestive Heart Failure, New York Heart Association (NYHA) IIIB or worse

Chronic renal failure (S-creatinine increased)

Immunosuppression (more than 10 mg daily of Prednisolone or stronger medication)

No axillary exploration planned

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2020-10-22 (Actual)

PRIMARY OUTCOMES:
Opiate consumption | 48 hours
  The cumulative consumption of opiates (Morphine). This is the most often used way to asses the efficacy of the regional anesthesia that the intervention consists of.
All cause mortality | 3 years and 5 years.
  This is to investigate the possible effect that a regional anesthesia may have on recurrence of a malignant tumor.

SECONDARY OUTCOMES:
Postoperative Nausea and Vomiting (PONV) | 48 hours
  PONV is common after general anesthesia and more so if opiates are used for analgesia. Measured on an ordinal scale 0=no PONV, 1=nausea, 2=vomiting, 3=repeated vomiting
Actual pain score | 48 hours
  To see if patients with a regional anesthesia have more or less pain than patients with intravenous Morphine as postoperative analgesia.
Recurrence of breast neoplasm | 3 and 5 years
  Recurrence of breast neoplasm
Chronic Pain | 6 (5-7) months after surgery
  Pain after 6 months as assessed in a telephone interview, measured as Numeric Rate Scale (0-10).

CONTACTS AND LOCATIONS:
Overall Officials: Joakim Johansson, PhD, Principal Investigator — Umea University
Locations (1):
- Östersund Hospital, Östersund, Jämtland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahlberg H, Wallgren D, Hultin M, Myrberg T, Johansson J. Less use of rescue morphine when a combined PSP/IPP-block is used for postoperative analgesia in breast cancer surgery: A randomised controlled trial. Eur J Anaesthesiol. 2023 Sep 1;40(9):636-642. doi: 10.1097/EJA.0000000000001795. Epub 2023 Jan 12. PMID 36633115